CLINICAL TRIAL: NCT01944527
Title: Cohort of Liver Transplanted Patients With Hepatitis C Virus Recurrence and Treated With Direct-acting Antiviral Agents
Brief Title: Use of Direct-acting Antiviral to Treat HCV Recurrence After Liver Transplantation (ANRSCO23CUPILT) Infection
Acronym: ANRSCO23CUPILT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013-A00941-44
Record Dates: First submitted 2013-09-13; First posted 2013-09-17 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: HCV Recurrence; Liver Transplantation; Direct-acting Antiviral Agents

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of direct-acting antivirals therapy in liver transplanted patients who experienced HCV recurrence.

This cohort is multicentric with constitution of biobank (plasma, serum) and the prospective collect of biological and clinical data's in the liver transplanted patients with recurrent HCV infection and treated with direct-acting anti-HCV agents.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years-old
* Liver transplanted patient
* Hepatitis C virus infection before transplantation
* HCV recurrence with a detectable HCV RNA before enrollment in cohort
* Use of at least one direct-acting antiviral agents with or without association with peginterferon and with or without association with ribavirin
* Treated by direct-acting antiviral agents or has been yet completed the treatment but still on follow up
* Affiliated to Health Insurance
* Written Signed consent form

Exclusion Criteria:

* Pregnant or breast-feeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant patients with recurrent hepatitis C virus infection treated with direct-acting antiviral agents and followed up in centers of transplantation of the university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 699 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The rate of sustained virological response 12 weeks after discontinuation of direct-acting anti-HCV therapy in liver transplanted patients with HCV recurrence | 12 weeks after discontinuation of therapy
  Sustained virological response (SVR) at 12 weeks after the end of the treatment (SVR defined as undetectable HCV RNA measured by PCR en real time at 12 weeks after antiviral therapy discontinuation)

SECONDARY OUTCOMES:
Virological responses at 1,2,3,4,6,8,12,16, 20, 24, 36, 48 weeks during treatment and 4,12,24,48 weeks after treatment discontinuation | Baseline, 1,2,3,4,6,8,12,16, 20, 24, 36, 48 weeks during treatement and 4,12,24,48 weeks after treatment discontinuation
  Detectability of HCV RNA according to real time PCR
Tolerability of direct acting antiviral HCV agents | Baseline, 1,2,3,4,6,8,12,16, 20, 24, 36, 48 weeks during treatment and 4,12,24,48 weeks after treatment discontinuation
  Clinical and laboratory parameters (hepatic, renal, hematological in particular) to assess safety and recording of adverse events
Drug-drug interactions | Baseline, 1,2,4,12,16, 24, 48 weeks during treatement and 4weeks after treatment discontinuation
  Trough blood concentration of immunosuppressive drugs
To evaluate emergence of viral resistance to direct-acting antivirals agents | Baseline, 1,2,3,4,6,8,12,16, 20, 24, 36, 48 weeks during treatement and 4,12,24,48 weeks after treatment discontinuation
To establish predictive factors of treatment failure and of emergence of viral resistance | Baseline, 1,2,3,4,6,8,12,16, 20, 24, 36, 48 weeks during treatement and 4,12,24,48 weeks after treatment discontinuation
  The rate of anticipated antiviral treatment discontinuation because of intolerability or of severe adverse events
Evaluate the incidence of graft loss and acute rejection | Day 0, 1,2,3,4,6,8,12,16, 20, 24, 36, 48 weeks during treatement and 4,12,24,48 weeks after treatment discontinuation
  The rate of graft loss
Impact on concomitant therapy on virological responses and safety | Baseline, 1,2,3,4,6,8,12,16, 20, 24, 36, 48 weeks during treatment and 4,12,24,48 weeks after treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Georges Philippe Pageaux, Professsor, Principal Investigator — HOSPITAL SAINT ELOI
Locations (1):
- Claire Fougerou, Rennes, France

REFERENCES:
- [Derived] Barrail-Tran A, Goldwirt L, Gele T, Laforest C, Lavenu A, Danjou H, Radenne S, Leroy V, Houssel-Debry P, Duvoux C, Kamar N, De Ledinghen V, Canva V, Conti F, Durand F, D'Alteroche L, Botta-Fridlund D, Moreno C, Cagnot C, Samuel D, Fougerou-Leurent C, Pageaux GP, Duclos-Vallee JC, Taburet AM, Coilly A. Comparison of the effect of direct-acting antiviral with and without ribavirin on cyclosporine and tacrolimus clearance values: results from the ANRS CO23 CUPILT cohort. Eur J Clin Pharmacol. 2019 Nov;75(11):1555-1563. doi: 10.1007/s00228-019-02725-x. Epub 2019 Aug 5. PMID 31384986
- [Derived] Antonini TM, Coilly A, Rossignol E, Fougerou-Leurent C, Dumortier J, Leroy V, Veislinger A, Radenne S, Botta-Fridlund D, Durand F, Houssel-Debry P, Kamar N, Canva V, Perre P, De Ledinghen V, Rohel A, Diallo A, Taburet AM, Samuel D, Pageaux GP, Duclos-Vallee JC; ANRS C023 CUPILT study group. Sofosbuvir-Based Regimens in HIV/HCV Coinfected Patients After Liver Transplantation: Results From the ANRS CO23 CUPILT Study. Transplantation. 2018 Jan;102(1):119-126. doi: 10.1097/TP.0000000000001928. PMID 28846559
- [Derived] Leroy V, Dumortier J, Coilly A, Sebagh M, Fougerou-Leurent C, Radenne S, Botta D, Durand F, Silvain C, Lebray P, Houssel-Debry P, Kamar N, D'Alteroche L, Petrov-Sanchez V, Diallo A, Pageaux GP, Duclos-Vallee JC; Agence Nationale de Recherches sur le SIDA et les Hepatites Virales CO23 Compassionate Use of Protease Inhibitors in Viral C in Liver Transplantation Study Group. Efficacy of Sofosbuvir and Daclatasvir in Patients With Fibrosing Cholestatic Hepatitis C After Liver Transplantation. Clin Gastroenterol Hepatol. 2015 Nov;13(11):1993-2001.e1-2. doi: 10.1016/j.cgh.2015.05.030. Epub 2015 Jun 1. PMID 26044317